CLINICAL TRIAL: NCT04686552
Title: Effects of Cinnamon Spice on Postprandial Glucose and Insulin in Normal Weight and Obese Individuals With Pre-Diabetes: A Pilot Study
Brief Title: Effect Cinnamon Spice on Postprandial Glucose and Insulin Responses
Acronym: CINNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18-000464
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Normal Weight; Overweight and Obesity
Keywords: cinnamon; insulin; glucose; postprandial; acute
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cinnamon (Experimental): The test meal consisted of ½ cup dry instant oatmeal, prepared with 1 cup of 2% milk served with 6 g of ground cinnamon.
  Interventions: Dietary Supplement: cinnamon
- control (No Intervention): The test meal consisted of ½ cup dry instant oatmeal, prepared with 1 cup of 2% milk served without 6 g of ground cinnamon

INTERVENTIONS:
Dietary Supplement: cinnamon — 6 g of ground cinnamon
  Other Names: control
  Arms: cinnamon

SUMMARY:
The objective of the proposed study is to investigate the effect of cinnamon on the postprandial glycemic response to a high glycemic index meal in normal and overweight/obese prediabetic subjects

DETAILED DESCRIPTION:
A randomized crossover study design will be carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins. There will be two groups of participants (normal and overweight/obese). Each participant will consume oatmeal prepared with 1 cup of 2% milk served with or without 6 g of ground cinnamon in random sequence. At each meal consumption blood will be collected to measure postprandial glucose and insulin at 0, 30, 60, 90, 120, 150 and 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adults age 20-50 years' old
* Typically consume low fiber/polyphenol diet (beige diet)
* normal weight individuals with a BMI of 18. to 24.9 kg/ m2 with fasting serum glucose <100 mg/dL
* overweight/obese individuals with a BMI of 25 to 35 kg/m2 and fasting serum glucose ≥100 mg/dL and <126 mg/dL or HbA1c >5.7% and < 6.5%.
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
* Any subject currently taking blood thinning medications such as Warfarin or Coumadin
* Any history of gastrointestinal disease or surgery except for appendectomy or cholecystectomy.
* Eating a high fiber/polyphenol diet or taking any medication or dietary supplement which interfere with the absorption of polyphenols.
* History of gastrointestinal surgery, diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP >95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history.
* Pregnant or breastfeeding
* Currently uses tobacco products.
* Currently has an alcohol intake > 20 g ⁄ day;
* Currently has a coffee intake > 3 cups ⁄ day;
* Allergy or sensitivity to cinnamon. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. To determine this, a positive history of cinnamon ingestion without incident will be requested. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
* Is lactose intolerant
* Is unable or unwilling to comply with the study protocol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
glucose | Baseline to 180 minutes
  postprandial glucose reponse
insulin | Baseline to 180 minutes
  postprandial insulin response

SECONDARY OUTCOMES:
C-peptide | Baseline to 180 minutes
  postprandial C-peptide response
glucagon | Baseline to 180 minutes
  postprandial glucagon reponse
lipids | Baseline to 180 minutes
  postprandial lipid response

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

REFERENCES:
- [Derived] Wang J, Wang S, Yang J, Henning SM, Ezzat-Zadeh Z, Woo SL, Qin T, Pan Y, Tseng CH, Heber D, Li Z. Acute Effects of Cinnamon Spice on Post-prandial Glucose and Insulin in Normal Weight and Overweight/Obese Subjects: A Pilot Study. Front Nutr. 2021 Jan 21;7:619782. doi: 10.3389/fnut.2020.619782. eCollection 2020. PMID 33553233